CLINICAL TRIAL: NCT02421757
Title: Treatment of Back Pain Using Transcutaneous Magnetic Stimulation (TCMS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Peter Rock, Professor of Anesthesiology, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00062233
Record Dates: First submitted 2015-04-10; First posted 2015-04-21 (Estimated); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-10

CONDITIONS: Lower Back Pain
Keywords: Transcutaneous Magnetic Stimulation; placebo
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Transcutaneous Magnetic Stimulation (Experimental): Transcutaneous Magnetic Stimulation
  Interventions: Device: Fischell Transcutaneous Magnetic Stimulation Pain Treatment Device
- Sham Device (Placebo Comparator): Sham Device
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Fischell Transcutaneous Magnetic Stimulation Pain Treatment Device — Transcutaneous Magnetic Stimulation
  Arms: Transcutaneous Magnetic Stimulation
Device: Placebo — The placebo Transcutaneous device
  Other Names: Fischell Transcutaneous Magnetic Stimulation Pain Treatment Device (TCMS Placebo)
  Arms: Sham Device

SUMMARY:
This is a single-site, randomized, Single-blinded, placebo-controlled, trial of Transcutaneous Magnetic Stimulation (TCMS) for the treatment of lower back pain. TCMS will be applied locally to the back in the location of a patient's pain.

DETAILED DESCRIPTION:
Approximately one third of Americans suffer from acute and chronic pain and pain has been called a silent epidemic. Treatment of pain often involves opioid medications with a significant potential for abuse, addiction and adverse reactions such as respiratory depression and death. Magnetic brain stimulation has been used for the treatment of pain. There are reports of its use in phantom-limb pain and in the treatment of central and peripheral pain syndromes.

The study will evaluate whether an experimental medical device (Fischell TCMS Pain Treatment Device) that emits pulses of a brief, intense magnetic field will relieve pain in the lower back. Transcutaneous Magnetic Stimulation (TCMS) is the name of this method of delivering magnetic pulses through the skin. TCMS has been approved by the FDA for peripheral nerve stimulation, treatment of migraine headaches and for depression but this type of device has not been studied scientifically for the treatment of back pain. No significant adverse reactions or side effects have been reported with the use of magnetic stimulation for headache treatment. Some patients who have migraine headaches have excellent pain relief with the magnetic treatment even if they do not get pain relief with medications. Other patients do not have headache relief with magnetic treatment. The current use of TCMS applied to the head requires special equipment and multiple treatment sessions. TCMS applied peripherally is easier to do, and may require fewer treatment sessions to achieve pain relief. Non-invasive treatment of pain would represent a significant advance in the field especially if its use both successfully treated pain and resulted in the reduction or elimination in the need for opioid medications.

The investigators do not know whether magnetic treatment will relieve back pain so the investigators will test this by applying a powerful electromagnet to the area of the back having pain. In some patients, the magnet will be turned on, but in other patients the magnet will not be turned on. Neither patients nor patient's treating doctor will know whether the magnet was turned on or not, although the study team will know which patients received treatment with magnetic pulses. The effect on pain will be recorded periodically for 2 days. If the patients' reported pain is reduced by having the magnet turned on compared to patients' who do not have the magnet turned on, then the magnet may have reduced the pain. Additional studies in patients will be needed to be sure that the magnet therapy is reducing low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, age >18 years of age
2. Prescription pharmacologic treatment is insufficient for treatment of pain
3. Pain duration of ≥ 6 months
4. Pain limits physical activity
5. Pain occurs daily
6. Chronic low back pain, with or without leg pain, associated with MRI or other imaging study consistent with lumbo-sacral spine disease with or without nerve compression
7. Pain intensity ≥ 5 at the time of enrollment a a self-reported pain score of ≥ 4 over the 7 preceding days.

Exclusion Criteria:

1. Life expectancy ≤ 6 months for any reason
2. Oral opiate dosing or type of opioid that has changed in past 12 months
3. Received intraspinal (e.g., epidural, intrathecal) medication in the past 6 months
4. Use of intravenous pain medication in the past 6 months
5. Active use of a transcutaneous electrical nerve stimulator (TENS) [within 30 days]
6. History of seizures
7. History of implanted medical device, cardiac pacemaker or implantable cardiac defibrillator, or other implant (Cochlear etc)
8. History of cardiac dysrhythmias
9. Member of vulnerable population
10. Current or potential legal action of disability claim related to back pain
11. Body Mass Index (BMI) >35
12. Another pain condition that might confound results, including back pain above the waistline
13. Women of child-bearing potential
14. Inability to undergo study assessments or complete questionnaires independently
15. Metal objects in the body (i.e. Aneurysm clip, bullet fragment)
16. Active psychological co-morbidites (i.e. uncontrolled schizophrenia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rock, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- La Toya Stubbs, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited at the Pain Management Center at University of Maryland Rehabilitation & Orthopaedic Institute from 8/22/2016-4/27/2017.
Pre-assignment Details: Patients who agreed to participate were provided with a pain diary and were instructed to document their average pain each day for a week using the Numeric Pain Rating Scale (NPRS) to establish their baseline level of pain. Patients were also given the Global Pain Scale (GPS) to complete and return on the day of treatment.
Period: Overall Study
Arm/Group | Transcutaneous Magnetic Stimulation | Sham Device
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcutaneous Magnetic Stimulation | Sham Device | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 7 | 16
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Immediate Pain Measured by Numeric Pain Rating Scale (NPRS)
Description: Immediate relief measured by Numeric Pain Rating Scale (NPRS)
  Scale from 0-10 0=No pain 10= Worse possible pain
Time Frame: 60 minutes
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Transcutaneous Magnetic Stimulation | Sham Device
Number analyzed (Participants) | 11 | 9
score on a scale | 4.89 [0 to 10] | 5.18 [0 to 10]

2. Secondary Outcome: Durable Pain Measured by Numeric Pain Rating Scale (NPRS)
Description: Durable pain relief measured by Numeric Pain Rating Scale (NPRS) 0= No pain 10= Worse imaginable pain
Time Frame: 30 days
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Transcutaneous Magnetic Stimulation | Sham Device
Number analyzed (Participants) | 11 | 9
score on a scale | 6.00 [0 to 10] | 6.57 [0 to 10]

ADVERSE EVENTS:
Time Frame: We collected information on adverse event data during the enrollment period of 30 days.
Description: This study had no risk of mortality
Arm/Group | Transcutaneous Magnetic Stimulation | Sham Device
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

LIMITATIONS AND CAVEATS:
The population of patients (chronic pain) proved to be difficult to get in for treatment and follow-up. This lead to small enrollment numbers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT02421757/Prot_SAP_000.pdf